CLINICAL TRIAL: NCT07234240
Title: Blinded Consumer Study for the Evaluation of the Usability and Efficacy of One Medical Device in Venous Return
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Millet Innovation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P023B24
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Venous Disease; Quality of Life; Symptoms and Signs
Keywords: Chronic venous disease; insoles; quality of life; symptoms; relief
MeSH Terms: conditions — Signs and Symptoms | interventions — Foot Orthoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: One medical device as investigational device (Experimental)
  Interventions: Device: Insoles

INTERVENTIONS:
Device: Insoles — Insoles At Day 0, the patient received the insoles and adapted them to his open shoes. The patient filled the quality-of-life's questionnaire at Day 0 and the same at Day14. The patient filled the rapid relief's questionnaire at Day7 and a usability's questionnaire at Day14.

SUMMARY:
The primary goal of this study was to assess, in vivo, the efficacy of the medical device Invisible insoles LIGHT LEGS in improving venous return in subjects affected by this problem after 14 days of medical device use, by self-assessment, filling in questions regarding Quality of Life, in comparison to the baseline.

The secondary goals of this study were (1) to assess in vivo the perception of subjects about the rapid relief felt after 7 days of using the same medical device, by selfassessment, filling-in three subjective evaluation questions, and (2) to assess in vivo the usability of the subjects regarding the same medical device after 14 days of its use, by self-assessment, filling in subjective evaluation questions.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Female/Male;
* Age: with 18 years old and older;
* Having signed an Informed Consent Form (ICF);
* Willingness, ability and likeliness to comply with all the study procedures and restrictions;
* Ability to give informed consent;
* Available during the entire study period;
* Understanding Portuguese language: Portuguese-speaking subjects capable of reading the documents;
* Affected by a symptomatic venous return problem;
* With a score >14 from the question 1 to 11 of the adapted CIVIQ questionnaire (each question scored on a scale from 0 to 4);
* Agree to wear open shoes suitable for insoles throughout the study, for at least 8 hours per day (with a heel <5cm);
* Having a shoe size of 36 to 41;

Exclusion Criteria:

* Known allergy or known history of hypersensitivity to the components of the investigational device and related compounds;
* Currently participating in another clinical study that may interfere with the study;
* Diagnosed skin diseases and/or cutaneous alterations on the test region (feet) that may impair the study (for example tattoos, marks, burns, scars, etc.);
* Diagnosed diseases that may impair the study (including but not limited to: Diabetes, Arteritis, Phlebitis, etc);
* Under pharmacological treatments on the 30 days previous to the beginning of the study and during the entire period of the study that may impair it (including but not limited to: inflammatory drugs, any drug that might cover the signs and symptoms, drugs with arterial or venous indications, etc.);
* Having applied any type of topical product (pharmaceutical, cosmetic or other) with similar effect of the medical device under study, on the test region (feet) during the study, besides the investigational device;
* Having a stage of CVD C3 on the CEAP classification;
* Having had a traumatic or neurological history in the last 6 months;
* Wearing an orthopaedic insole made by a health professional;
* Having a significant and disabling lower limb pain;
* Having a significant and disabling back pain;
* Having a contraindication to wearing insoles and open shoes;
* Wearing open shoes with an anatomical shape (e.g. Birkenstock);
* Pregnancy or intention to conceive during the study;
* Breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Day 0 and Day 14
  CIVIQ (ChronIc Venous Insufficiency Quality of Life Questionnaire) 20 : It is a quality of life assessment scale comprising 20 items grouped into four main dimensions (pain, physical, psychological, social) with 5 levels (0 point (min) to 4 points (max)).The final score is between 0 and 80 points. A low score indicates a low impact of the disease on quality of life.

SECONDARY OUTCOMES:
Rapid relief | Day 7
  Perception of subjects about the rapid relief felt after 7 days (t7) of using the medical device, by self-assessment, filling-in three subjective evaluation questions
Usability evaluation | Day 14
  Usability of the subjects regarding the same device, through subjective evaluation questions filled by the subjects after 14 days (D14) of using the medical device.

CONTACTS AND LOCATIONS:
Locations (1):
- Juliana Gouveia, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No